CLINICAL TRIAL: NCT02079142
Title: Implementation of Evidence-based Treatments for On-campus Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Denise Wilfley, Principal Investigator, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R01MH095748-01 (NIH); 1R01MH095748 (NIH)
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Eating Disorders (Excluding Anorexia Nervosa); Depression
MeSH Terms: conditions — Feeding and Eating Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Intensity Strategy: Train-the-trainer (Experimental): One therapist from each counseling center randomized to this arm will be selected to become the trainer and will be trained to train their colleagues.
  Interventions: Behavioral: High Intensity Strategy: Train-the-trainer
- Low Intensity Strategy: Expert Consultation (Active Comparator): The IPT expert from Washington University will travel to all counseling centers randomized to this condition and train all participating therapists on site and be available for monthly phone consultation for up to one year following training on site.
  Interventions: Behavioral: Low Intensity Strategy: Expert Consultation

INTERVENTIONS:
Behavioral: High Intensity Strategy: Train-the-trainer — Trainers in the high intensity condition will attend two separate workshops at Washington University in St. Louis designed to teach participants to conduct IPT and then to train IPT. Following participation in the first, two-day workshop, each trainer will return to their site and be encouraged to treat at least two cases with eating disorders or depression, audio recording each session.
  Trainers will then return to Washington University to be trained in how to train their other staff members in IPT.
  Arms: High Intensity Strategy: Train-the-trainer
Behavioral: Low Intensity Strategy: Expert Consultation — Investigators will provide a two-day workshop on IPT at each site randomized to this condition to train therapists to use IPT for the treatment of Eating Disorders and depression.
  Arms: Low Intensity Strategy: Expert Consultation

SUMMARY:
The purpose of this study is to evaluate two training methods of IPT with mental health service providers in college counseling centers.

DETAILED DESCRIPTION:
Although there have been major advances in developing evidence-based psychotherapies, the adoption of such treatments by community therapists has been slow. One of the problems is the difficulty therapists in practice have in learning how to conduct an evidence-based psychotherapy. Hence, this study will investigate two methods of teaching therapists interpersonal therapy (IPT), an evidence based treatment for eating disorders and depression, at 40 college or University counseling centers.

Current approaches to training therapists to conduct new treatments typically consist of a one or two day workshop delivered by an expert and provision of a manual for the therapy in question. Recent reviews have concluded that while workshops increase therapists' knowledge, their impact on skills may be short-lived without further consultation. Thus, investigators will supplement IPT training manuals and workshops by offering monthly consultation calls to participating therapists for 12 months following the workshop. The consultation calls are not designed to be case supervision per se. Rather, they are to be seen as extended training on IPT. This training condition is referred to as expert consultation.

The second training strategy, referred to as train-the-trainer, features expertise capacity building within each organization. There is a strong theoretical case for this implementation strategy as it is based on the principles of social cognitive theory, featuring active learning via modeling, feedback on performance, building self-efficacy, and supportive interactions among therapists developing IPT skills. This 'train-the-trainer' approach involves active learning which centers around development of an internal coach and champion, and has been recommended as the most effective means of changing actual therapist behaviors rather than just attitudes and self-reported proficiency. Roth et al. have made the case that effective implementation of evidence-based treatment in routine clinical services requires that the training approximate that which characterized the research context (e.g., continuing feedback and supervision and monitoring of treatment fidelity). Our train-the-trainer strategy offers a practical means of accomplishing this goal.

ELIGIBILITY:
Inclusion Criteria:

* Currently employed in a participating university counseling center
* Providing regular student-client services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2012-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Treatment Fidelity | up to 53 months
  Treatment fidelity comprises two dimensions: adherence to the procedures of IPT and level of competence in applying these procedures.

SECONDARY OUTCOMES:
Student Symptom | up to 53 months
  Eating Disorder and Depression psychopathology will be assessed using a separate count of binge eating and purging (including episodes of self-induced vomiting, episodes of laxative and diuretic use, and episodes of fasting defined as 24 hours without food) for eating disorders and the PHQ-9 for Depression. This measure correlates well with data obtained from structured interviews. This measure will allow us to test the relationship between fidelity to IPT and client outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Denise E Wilfley, Ph.D., Principal Investigator — Washington University School of Medicine; Stewart Agras, MD, Principal Investigator — Stanford University; Terrance G Wilson, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Derived] Raghavan R, Fitzsimmons-Craft EE, Welch RR, Jo B, Proctor EK, Wilson GT, Agras WS, Wilfley DE. Cost-effectiveness of train-the-trainer versus expert consultation training models for implementing interpersonal psychotherapy in college mental health settings: evidence from a national cluster randomized trial. Implement Sci. 2024 Jul 29;19(1):55. doi: 10.1186/s13012-024-01388-2. PMID 39075590
- [Derived] Wilfley DE, Agras WS, Fitzsimmons-Craft EE, Bohon C, Eichen DM, Welch RR, Jo B, Raghavan R, Proctor EK, Wilson GT. Training Models for Implementing Evidence-Based Psychological Treatment: A Cluster-Randomized Trial in College Counseling Centers. JAMA Psychiatry. 2020 Feb 1;77(2):139-147. doi: 10.1001/jamapsychiatry.2019.3483. PMID 31693069